CLINICAL TRIAL: NCT06815796
Title: Loop Vs. Anchor Tenodesis of the Long Head of the Biceps Brachii Tendon. a Prospective, Randomized, Double-blinded Study
Brief Title: Loop Vs. Anchor Tenodesis of the Long Head of the Biceps Brachii Tendon
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Krankenhaus Barmherzige Schwestern Linz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EK 1249/2022
Record Dates: First submitted 2024-12-01; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Biceps Tendon Disorder; Shoulder Arthroscopic Surgery
Keywords: Biceps Tendon Pathology; Arthroscopic Tenodesis; Loop Tenodesis; Suture Anchor Tenodesis; Clinical outcomes; Return to sport

STUDY DESIGN:
Intervention Model Description: Randomized allocation to 2 groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Loop tenodesis of Long head of biceps tendon (Experimental): Long head of biceps tenodesis using loop technique
  Interventions: Procedure: Arthroscopic Loop tenodesis of long head of biceps.
- Anchor tenodesis of Long head of biceps tendon (Active Comparator): Long head of biceps tenodesis using anchor technique
  Interventions: Procedure: Anchor Tenodesis of Long head of biceps tendon

INTERVENTIONS:
Procedure: Arthroscopic Loop tenodesis of long head of biceps. — Loop tenodesis of the long head of biceps tendon.
  Arms: Loop tenodesis of Long head of biceps tendon
Procedure: Anchor Tenodesis of Long head of biceps tendon — Anchor Tenodesis of Long head of biceps tendon
  Arms: Anchor tenodesis of Long head of biceps tendon

SUMMARY:
The goal of this clinical trial is to learn if loop tenodesis is as effective as suture anchor tenodesis for treating long head of biceps (LHB) pathology. It will also assess the safety and outcomes of both techniques. The main questions it aims to answer are:

How effective is loop tenodesis compared to suture anchor tenodesis in preventing shoulder deformities and maintaining biomechanical strength? What complications or failures occur with each technique? Researchers will compare suture anchor tenodesis using the Arthrex FiberTak system with loop tenodesis (an implant-free technique).

Participants will:

Undergo surgery with either suture anchor tenodesis or loop tenodesis, assigned randomly.

Be informed about the procedure and sign a consent form prior to surgery. Have their clinical outcomes evaluated and compared before and after their treatment.

DETAILED DESCRIPTION:
A pathology of the long head of the biceps tendon (LHB) is often the cause of shoulder pain. There are numerous ways to treat an LHB pathology. Arthroscopic biceps tenotomy is a simple method to address this condition. However, it often results in a cosmetic "Popeye deformity" and reduced strength during abduction. For this reason, and due to advancements in anchor systems, arthroscopic biceps tenodesis using an anchor in the bicipital groove is becoming increasingly popular. The advantage of this method is that it prevents potential muscle deformity and provides stable fixation in the bicipital groove. Possible disadvantages include potential failure and the cost of the anchors used.

A newer method with good biomechanical and clinical outcomes is the so-called arthroscopic loop tenodesis. In this technique, the LHB is proximally detached at its insertion and shuttled extracapsularly using a clamp. The end of the tendon is then folded and sutured into a so-called "loop." The tendon is released, and after spontaneous retraction, it forms a so-called autotenodesis in the bicipital groove. This technique has the advantage of providing implant-free fixation while also demonstrating good biomechanical outcomes.

The goal of this study is to investigate and compare the clinical success rate after arthroscopic treatment of the LHB using either a suture anchor tenodesis (Arthrex FiberTak) or the so-called loop tenodesis (implant-free fixation). The study is being conducted in the Orthopedics Department of the Ordensklinikum Linz - Barmherzige Schwestern, Austria.

All patients requiring arthroscopic biceps tenodesis at the Orthopedics Department of the Ordensklinikum Linz will be treated using either suture anchor tenodesis or loop tenodesis. Allocation to the surgical technique will be determined by block randomization (block length = 9) immediately after the decision to include the patient in the study. Block randomization using a random number generator is chosen to ensure that the group sizes are approximately equal.

Before surgery, patients will be informed about the study process and the possibility of participation during a personal consultation. They will also receive a patient information and consent form in which their agreement to participate is documented in writing. Patients will receive a copy of the signed consent form, while the original remains with the investigator.

The data collected in this study will be analyzed individually and compared with existing data in the literature. The results will then be taken into account when considering various treatment concepts, potentially leading to adjustments or optimizations to benefit the patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring a tenodesis of the long head of the biceps tendon during the study period, using either anchor tenodesis or loop tenodesis.
* Patients must be at least 18 years old.
* Patients must have the capacity to give informed consent.

Exclusion Criteria:

* Patients with insufficient documentation.
* Patients under the age of 18.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley Score | up to 24 months
  score ranges from 0 to 100 points, representing worst and best shoulder function
American Shoulder and Elbow Surgeons score (ASES) | up to 24 months
  ranges from 0 to 100, with 0 the lowest level of function and 100 the highest level of function
Disabilities of the arm, shoulder and hand (DASH) outcome questionnaire | up to 24 months
  scored 0 (no disability) to 100

SECONDARY OUTCOMES:
Cosmetic Outcome | up to 24 months
  Incidence of "Popeye deformity" post-surgery
Strength | up to 24 months
  Supination of the forearm in 90 degree elbow flexion in kilogram
Complications | up to 24 months
  Rate of complications (anchor failure, Pop-eye deformity, infections, pain etc.)
Pain (pre-/postOP) | up to 24 months
  assessed using a Visual Analog Scale (VAS). two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Sport activities | up to 24 months
  assessed using a questionnaire
Level of sport | up to 24 months
  assessed using a questionnaire (amateur (no salary), professional (salary)
Sport duration | up to 24 months
  assessed using a questionnaire (1x/2x/3x/4x/>4x per week; 0-15 min, 16-30 min, 31-60 min, 61-120 min, > 120 min per day)
Return to sport | up to 24 months
  assessed using a questionnaire (months)
Pain during sport | up to 24 months
  assessed using a questionnaire with virtual analag scale (pre- and postOP; VAS 0-10, 0= no pain, 10= maximal pain)
Fear during sport | up to 24 months
  assessed using a questionnaire with virtual analog scale (pre- and postOP; VAS 0-10, 0= no fear, 10= maximal fear)

CONTACTS AND LOCATIONS:
Locations (1):
- Ordensklinikum Linz Barmherzige Schwestern, Linz, Austria

IPD SHARING:
Plan to Share IPD: No
IPD can be shared upon request, due to government privacy policy routine uploading of specific data can not be done.